CLINICAL TRIAL: NCT00379197
Title: Phase II Study of Naltrexone for the Treatment of Hormone-Refractory, Metastatic Breast Cancer
Brief Title: Phase II of Naltrexone in Hormone-Refractory Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006LS016; UMN-0604M85308 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer, estrogen receptor positive; recurrent breast cancer; hormone-refractory, metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Naltrexone; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Naltrexone (Experimental): Naltrexone 50 mg will be taken orally once a day every day of a 28 day treatment course (cycle 1) and continue for another identical 28 day treatment (cycle 2) . PET scan will be performed after cycle 1 and cycle 2 complete.
  Interventions: Drug: naltrexone; Procedure: PET scan

INTERVENTIONS:
Drug: naltrexone — Naltrexone 50 mg will be orally taken once daily for 28 day (cycle 1), and continues once daily for another 28 days (cycle 2) without interval.
  Other Names: REVIA
Procedure: PET scan — Patients will receive PET scan approximately one hour after being injected with 2-Deoxy-2-[18F]fluoro-D-Glucose (FDG). PET scans will be performed after the completion of cycle 1 and cycle 2 and during the 1 year follow-up.
  Other Names: Positron-emission tomography scan

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Naltrexone may fight breast cancer by blocking the use of estrogen by the tumor cells. Naltrexone may also stop the growth of breast cancer by impairing blood flow to the tumor.

PURPOSE: This phase II trial is studying how well naltrexone works in treating women with metastatic breast cancer that is no longer responsive to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of naltrexone in women with hormone-refractory, metastatic breast cancer as measured by serial fludeoxyglucose F 18 positron emission tomography-CT scans.

Secondary

* Determine the safety of naltrexone in these patients.
* Determine the median time to event (first time when maximum specific uptake values is higher than that at baseline) within 1 year of study entry.

OUTLINE: This is an open-label study.

Patients receive oral naltrexone once daily for 8 weeks in the absence of disease progression or unacceptable toxicity. After 8 weeks, patients may continue naltrexone off study at the discretion of the physician.

Patients undergo fludeoxyglucose F 18 positron emission tomography-CT scans at baseline, week 4, week 8, and periodically thereafter.

After completion of study treatment, patients are followed for up to 1 year.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, hormone-receptor positive breast cancer
* Disease that has progressed despite previous systemic hormonal therapy. Hormone therapy must be terminated at least 2 weeks prior to study enrollment.
* Prior chemotherapy, immunotherapy, or biological therapy is allowed if at least 3 weeks since last treatment. Patient must recover from the acute toxic effects of the treatment prior to study enrollment.
* Measurable disease as defined by solid tumor response (RECIST) criteria or non-measurable bone disease that is Positron-emission tomography (PET) avid
* Karnofsky performance status >70%
* Female, age 18 years or older
* Adequate organ function within 14 days of study enrollment including the following:

  * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 10^9/L, platelets >75 x 10^9/L, and hemoglobin > 8 g/dL
  * Hepatic: bilirubin ≤ 2 times the upper limit of normal (× ULN), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2 × ULN. (AST and ALT ≤ 5 × ULN is acceptable if liver has tumor involvement)
  * Renal: creatinine ≤ 2 times the upper limit of normal
* Women of childbearing potential are required to use an effective method of contraception (ie, a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study and for 3 months after the last dose of study drug.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion criteria:

* Brain metastases unless stable for 1 month or more following radiation therapy.
* Pregnant or lactating women. PET-CT is not approved during pregnancy. A negative urine or serum pregnancy test is required for all females of child bearing potential within 7 days prior to study entry. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Use of any short-acting or long-acting opioid medication (including morphine, meperidine, oxycodone, hydromorphone, hydrocodone, fentanyl, tramadol) within 10 days prior to study enrollment
* Pain uncontrolled with the use of non-narcotic drugs (acetaminophen or non-steroidal medications)
* History of sensitivity to naltrexone
* Acute hepatitis or liver failure
* Immunosuppressive therapy for patients with autoimmune diseases, organ transplant, or other indications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Yee, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Vijayakumar J, Haddad T, Gupta K, Sauers J, Yee D. An open label phase II study of safety and clinical activity of naltrexone for treatment of hormone refractory metastatic breast cancer. Invest New Drugs. 2023 Feb;41(1):70-75. doi: 10.1007/s10637-022-01317-4. Epub 2022 Nov 28. PMID 36441436

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone: Naltrexone 50 mg taken orally once daily for 2 28-day cycles with an option to continue on Naltrexone at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Naltrexone
Started | 13
Completed | 8
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Naltrexone: Naltrexone hydrochloride 50 mg will be taken once a day every day of a 28 day treatment course. Positron-emission tomography (PET) / computed tomography (CT) given with injection of 2-Deoxy-2-[18F]fluoro-D-Glucose (FDG).
  naltrexone hydrochloride: Naltrexone should be taken with water or food, and it can be taken at any time day. Naltrexone 50 mg will be taken once a day every day of a 28 day treatment course.
  Positron-emission tomography (PET) / computed tomography (CT): Given with injection of 2-Deoxy-2-[18F]fluoro-D-Glucose (FDG). Follow-up scans will be performed after the completion of cycle 1 and cycle 2 and during the 1 year follow-up.
Arm/Group | Naltrexone
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Sex/Gender, Customized [Number; unit: participants]
  Female only | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Disease Response
Description: A response is the number of participants whose tumor demonstrated a decrease in FDG uptake (SUV) by 50% or greater in at least one of the metastatic sites as measured by PET imaging at the end of 4 weeks of treatment compared to baseline.
Time Frame: Week 4
Measure: Number; unit: participants
Groups:
- Naltrexone Treatment: Naltrexone 50 mg will be orally taken once daily for 28 day (cycle 1), and continues once daily for another 28 days (cycle 2) without interval. PET scan will be performed as baseline level at the beginning of study and after the completion of cycle 1 and cycle 2.
Arm/Group | Naltrexone Treatment
Number analyzed (Participants) | 8
participants | 1

2. Secondary Outcome: Median Time to Event
Description: First time when maximum SUV is higher than that at baseline within 1 year of study entry.
Time Frame: From Baseline to 1 Year
Population: One of the 8 participants did not have an increase in SUV above baseline at 8 weeks, but no further PET scans were performed after 8 weeks. The reported median value is for the remaining 7 participants.
Measure: Median (Full Range); unit: weeks
Arm/Group | Naltrexone
Number analyzed (Participants) | 7
weeks | 8 [4 to 8]

ADVERSE EVENTS:
Groups:
- Naltrexone Treatment: Naltrexone 50 mg will be orally taken once daily for 28 day (cycle 1), and continues once daily for another 28 days (cycle 2) without interval. PET scan will be performed after the completion of cycle 1 and cycle 2 and during the 1 year follow-up compared to the baseline level of FDG uptake.
Arm/Group | Naltrexone Treatment
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone Treatment (N=8)
Anemia (Blood and lymphatic system disorders) | 1
Pain right axillary node (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Abdominal bloating (Gastrointestinal disorders) | 1
right upper quadrant abdominal pain (Gastrointestinal disorders) | 1
increased thirst (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Cirrhotic Appearing Liver (Hepatobiliary disorders) | 1
Weight Gain (Investigations) | 1
pain - muscular (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Psychiatric disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
mild erythema (Skin and subcutaneous tissue disorders) | 1
hand and foot syndrome (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes